CLINICAL TRIAL: NCT06507527
Title: ASSESSMENT OF THE ADEQUACY IN CARE OF THE FRAGILE PATIENT IN A DIGESTIVE ENDOSCOPY UNIT FRIEND Study (FRailty In ENDoscopy) Estudi FRIEND (FRailty In ENDoscopy)
Brief Title: Frailty in Outpatient Digestive Endoscopy
Acronym: FRIEND
Status: Recruiting | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Other Study IDs: FRIEND
Record Dates: First submitted 2024-06-18; First posted 2024-07-18 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Frailty; Comorbidities and Coexisting Conditions; Complication
Keywords: Endoscopy; Indication; Bowell Preparation; Adverse effects
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Outpatients over 70 years of age referred to the Digestive Endoscopy Unit: Collection of variables: demographic variables, comorbidity, frailty (specific questionnaires), digestive endoscopy (upper and/or lower), possible complications related to the endoscopic process and the profitability and impact of the endoscopy.
  Interventions: Other: Collection of variables

INTERVENTIONS:
Other: Collection of variables — This is an observational study, so no interventions that are not routine clinical practice are performed. It is only about collecting information on variables that are already collected in normal clinical practice.

SUMMARY:
The increase in our society of the proportion of frail people who suffer from disability and dependency forces us to detect modifiable factors and therefore subject to intervention that can adapt health care for frail patients in order to increase the effectiveness and safety of medical treatments and procedures.

A geriatric assessment should be performed on all patients likely to present frailty prior to a digestive endoscopy to assess the risk-benefit of the indication and to improve patient preparation by avoiding adverse effects of endoscopic examinations, increasing the safety and profitability of the tests There are no data in our medium on the prevalence of frailty in patients referred for endoscopy, nor on the incidence in these patients of adverse effects, inadequate preparations, or incomplete examinations, so a frailty study is needed to elaborate multidisciplinary protocols that improve circuits and care in these patients and prevent complications.

The questions we want to try to answer are:

* Prevalence and severity of fragility in digestive endoscopy.
* Specific problems related to fragility in digestive endoscopy, mainly the profitability of the examination and the incidence of adverse effects, in order to create protocols for improving care in this group of patients.

DETAILED DESCRIPTION:
This is a prospective observational study.

In all patients older than 70 years referred for an ambulatory endoscopy, the presence of frailty and its degree will be assessed through validated questionnaires commonly used in the preparation of the patient for digestive endoscopy. A nurse trained by the Geriatrics Service of our hospital carries out a telephone contact with the patient or the patient's caregiver to fill out the questionnaires.

The formation of subgroups of patients will be assessed for the statistical analysis in relation to the degree of frailty and the type of endoscopy (upper or lower digestive endoscopy)

A random sample of 1474 individuals is sufficient to estimate, with 95% confidence and an accuracy of +/- 2.5 percentage units, a prevalence of frailty in the study population that is expected to be around 40%. Given that at this stage it is a cross-sectional study, no follow-up losses are expected.

Since the main aim of the study is cross-sectional, it is necessary to estimate the prevalence of frailty and a 95% confidence interval calculated using an exact method (Clopper-Pearson method).

The analysis of the profitability of the indication and of the adverse effects, as outcomes of interest in the achievement of the secondary objectives, will be analyzed according to the degree of frailty (main factor of the study). Likewise, the effect of potentially confounding variables will be studied, on the degree of fragility, and also on each of the outcomes taken into consideration. Finally, a multivariate analysis for each outcome will be used to evaluate the possible causal association with the degree of frailty, adjusting in each analysis for potentially confounding variables.

For the analyzes the statistical package STATA 15.1 and R will be used in the version that is updated at the time of the statistical analysis.

Basic patient demographic data (age, sex) will be collected. The presence of multipathology will be assessed using the CIRS(G)-Charlson questionnaire. Data related to the patient's frailty will be collected using the CFS and FRAGIL-VIG questionnaires.

Information about the endoscopic procedure will be collected with data recorded in the medical history. The cleaning agent and the degree of compliance with the colon cleaning protocol (diet, fasting, volume ingested, fractionation of the cleaning agent) will be noted in the clinical history, as well as the incidents that occurred in relation to the preparation for endoscopy.

In the endoscopic report, data on the preparation of the colon and intra-trial complications will be recorded.

Information on post-test complications will be collected with the data recorded in the clinical record. Only relevant adverse effects that require medical attention will be recorded, not considering minor adverse effects because they are not relevant to our study, since they do not provide information that helps to improve the care of the fragile patient in the field of endoscopy.

Frailty is defined as a CFS rating greater than 4 or a FRAGIL-VIG value greater than 0.

Adequate preparation is defined as a Boston Cleansing Classification rating of 2 or 3 in each and every segment of the colon.

The endoscopy indication is defined as unprofitable in the following cases:

* The patient does not show up or reschedules the examination
* The patient appears but it is not possible to perform the examination due to decompensation of the underlying pathology or for not having been able to comply with the test preparation protocols.
* The patient appears and the endoscopic examination is carried out, but it is not possible to give an adequate diagnosis or to carry out a therapeutic under safe conditions.

The cost-effectiveness calculation will be done by calculating the overall percentage of patients in which there are no situations that prevent an adequate diagnosis and/or therapy, and the causes of lack of cost-effectiveness will be calculated based on the assumptions explained in the text.The calculation of the cost of the endoscopy indication is closely related to the concept of profitability. All cases with a lack of profitability conceptually maintain the indication of the test and therefore need repetition of their request, given that the diagnostic-therapeutic objective of the initial indication has not been achieved. The cost of the hypothetical repetition of these scans will be calculated based on the prices established for each type of endoscopy and a cost comparison will be made between the different degrees of fragility.

A relevant adverse effect is defined in the following cases:

* Decompensation of underlying pathology that requires hospital care
* Complications related to sedation
* Post-colonoscopy bleeding
* Post-colonoscopy perforation

ELIGIBILITY:
Inclusion Criteria:

* It will include all patients over 70 years of age who are indicated to undergo an ambulatory upper or lower endoscopy.

Exclusion Criteria:

* Age below 70 years
* Non-ambulatory endoscopies
* Assessment of test contraindications by the endoscopist
* Non-acceptance to enter the study

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Outpatients may be referred from hospital consultations or from out-of-hospital medical centers. Age is the inclusion criterion so that frailty can be assessed in patients over 70 years of age, who are the patients with the highest risk of presenting a frailty condition.
Sampling Method: Probability Sample
Enrollment: 1474 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of frailty | At the moment of telephone contact with the patient
  Valuated frailty questionnaires (CFS and FRAGIL-VIG). Frailty is defined as a CFS rating greater than 4 or a FRAGIL-VIG value greater than 0. The degree of frailty is determined by FRAGIL-VIG score. The frailty questionnaires are completed during nurse telephone contact with the patient, prior to the digestive endoscopy.

SECONDARY OUTCOMES:
Profitability of the endoscopy indication. | At the moment of endoscopy.
  The endoscopy indication is defined as unprofitable in the following cases:
  * The patient does not show up or reschedules the examination
  * The patient appears but it is not possible to perform the examination due to decompensation of the underlying pathology or for not having been able to comply with the test preparation protocols.
  * The patient appears and the endoscopic examination is carried out, but it is not possible to give an adequate diagnosis or to carry out a therapeutic under safe conditions.
  The profitability calculation will be done by calculating the overall percentage of patients in which there are no situations that prevent a diagnosis and/or adequate therapy
Cost of the endoscopy indication | At the moment of endoscopy
  The calculation of the cost of the endoscopy indication is closely related to the concept of profitability. All cases with a lack of profitability conceptually maintain the indication of the test and therefore need repetition of their request, given that the diagnostic-therapeutic objective of the initial indication has not been achieved. The cost of the hypothetical repetition of these scans will be calculated based on the prices established for each type of endoscopy and a cost comparison will be made between the different degrees of fragility.
Incidence of relevant complications during the endoscopy process. | 30 days after digestive endoscopy.
  A relevant adverse effect is defined in the following cases:
  * Decompensation of underlying pathology that requires hospital care
  * Complications related to sedation
  * Post-colonoscopy bleeding
  * Post-colonoscopy perforation
  The patient's medical history will be reviewed 30 days after the endoscopy to collect data on possible relevant complications.
Clinical impact of the endoscopy indication | Up to 2 months after endoscopy
  The clinical impact will be measured based on whether the endoscopy performed leads to:
  * Absence of information in relation to the medical process investigated
  * A clinical diagnosis in relation to the medical process investigated
  * A clinical diagnosis not related to the medical process investigated
  * A therapeutic intervention After the clinical evaluation and medical decision on the result of the endoscopy by the requesting doctor or the endoscopist
Degree of frailty | At the moment of telephone contact with the patient
  The degree of frailty is determined by FRAGIL-VIG score (<0,20 absence of frailty or pre-frailty, 0,20-0,35 initial, 0,36-0,50 intermediate, >0,50 advanced)

CONTACTS AND LOCATIONS:
Overall Officials: AGUSTIN SEOANE URGORRI, MD, Principal Investigator — Parc de Salut Mar. Hospital del Mar
Locations (1):
- Parc de Salut Mar. Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All data collected will be entered into a database so that statistical analysis can later be carried out. This database must subsequently be shared with the statistics service of our hospital in order to perform an appropriate statistical analysis.
Supporting Information: SAP
Time Frame: Once patient recruitment is completed, the statistician will have the study data available for as long as he or she considers appropriate to perform the analyses. The time required until the study is accepted for publication is considered appropriate.
Access Criteria: The statistician will have access to the entire study database for the relevant statistical analyses.

REFERENCES:
- [Background] Machlab S, Francia E, Mascort J, Garcia-Iglesias P, Mendive JM, Riba F, Guarner-Argente C, Solanes M, Ortiz J, Calvet X. Risks, indications and technical aspects of colonoscopy in elderly or frail patients. Position paper of the Societat Catalana de Digestologia, the Societat Catalana de Geriatria i Gerontologia and the Societat Catalana de Medicina de Familia i Comunitaria. Gastroenterol Hepatol. 2024 Jan;47(1):107-117. doi: 10.1016/j.gastrohep.2023.05.004. Epub 2023 May 18. English, Spanish. PMID 37209916
- [Background] Oberndorfer T, Jurawan R. Frailty should be assessed in older patients considered for colonoscopy. N Z Med J. 2021 Jul 30;134(1539):74-76. No abstract available. PMID 34320617
- [Background] Cha JM, Kozarek RA, La Selva D, Gluck M, Ross A, Chiorean M, Koch J, Lin OS. Risks and Benefits of Colonoscopy in Patients 90 Years or Older, Compared With Younger Patients. Clin Gastroenterol Hepatol. 2016 Jan;14(1):80-6.e1. doi: 10.1016/j.cgh.2015.06.036. Epub 2015 Jul 9. PMID 26164224
- [Background] Taleban S, Toosizadeh N, Junna S, Golden T, Ghazala S, Wadeea R, Tirambulo C, Mohler J. Frailty Assessment Predicts Acute Outcomes in Patients Undergoing Screening Colonoscopy. Dig Dis Sci. 2018 Dec;63(12):3272-3280. doi: 10.1007/s10620-018-5129-x. Epub 2018 May 24. PMID 29796910
- See also: World report on aging and health. [Internet]. Geneva: World Health Organization.2015 — http://apps.who.int/iris/bitstream/10665/186466/1/9789240694873_spa.pdf
- See also: Population Projections 2018 [Internet]. Statistics National Institute; 2018 — http://www.ine.es/prensa/pp_2018_2068.pdf